CLINICAL TRIAL: NCT00536107
Title: A Randomized/Open Label/Parallel Group/Multicenter/Phase IV Study to Assess Safety/Tolerability/Efficacy of Oral Gefitinib 250 mg Versus IV Docetaxel 60 mg/m2 in Patients With Locally Advanced or Metastatic NSCL Cancer of Adenocarcinoma Histology Previous Treated With One Platinum Base Chemotherapy
Brief Title: Study to Assess Safety/Tolerability/Efficacy of Gefitinib Versus Docetaxel in Locally Advanced or Metastatic Non-Small Cell Lung Cancer (NSCLC)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D7913C00046
Record Dates: First submitted 2007-09-26; First posted 2007-09-27 (Estimated); Results first posted 2013-10-01 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-08

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Non-Small Cell Lung Cancer; Locally Advanced or Metastatic NSCL Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib; Magnetic Resonance Spectroscopy; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Docetaxel (Active Comparator): docetaxel
  Interventions: Procedure: CT or MRI; Drug: Docetaxel
- Gefitinib (Experimental): Gefitinib (IRESSA)
  Interventions: Drug: Gefitinib; Procedure: CT or MRI

INTERVENTIONS:
Drug: Gefitinib — 250 mg oral
  Other Names: IRESSA
  Arms: Gefitinib
Procedure: CT or MRI — performed at screening and every 6 weeks
Drug: Docetaxel — 60mg/m2 intravenous infusion
  Other Names: Paxel
  Arms: Docetaxel

SUMMARY:
This is a randomized, open- label, parallel group, phase IV, multicentre study. The total number of patients expected to be recruited is 40. These randomized patients will have a histologically or cytologically confirmed adenocarcinoma histology of locally advanced or metastatic NSCLC. Patients will be recruited by investigational sites that have expertise in treating patients with non-small cell lung cancer. The study will compare gefitinib monotherapy 250 mg/day orally with docetaxel 60 mg/m2 intravenously over 1 hour every 3 weeks with a primary endpoint of safety and tolerability. The target population will be patients who have received one prior platinum-based chemotherapy and are now considered suitable candidates for further chemotherapy with docetaxel. At study entry, patients will be randomized on a 1:1 basis stratified with respect to performance status (0-1 vs. 2). Patients may continue to receive treatment with either gefitinib or docetaxel until disease progression, unacceptable toxicity or the occurrence of any of the other specific criteria. An independent committee will be appointed to perform a blinded review of all patient scans. Any assessments/visits after screening should be performed within a window of plus or minus 3 working days of the scheduled visit date. If selected screening evaluations are done within 7 days of Day 1, Cycle 1 of treatment, and are acceptable for study entry, they do not have to be repeated on Day 1 unless the investigator believes that they are likely to have significantly changed. Any patient who discontinues from study treatment without radiological evidence of disease progression (except for withdrawal of consent by patient) should continue to have objective tumor assessments every 6 weeks in order to collect information on progression of disease

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced (Stage IIIB) or metastatic (Stage IV) NSCLC, not amenable to curative surgery or radiotherapy
* Treatment with one prior chemotherapy regimen, which must have been platinum based* *Patients must have demonstrated radiological or clinical progression since completion of previous chemotherapy regimen.
* Adequate hepatic function, defined as BOTH a bilirubin < upper limit of reference range (ULRR) AND an "Eligible" combination of transaminases (aspartate aminotransferase (AST) or alanine aminotransferase (ALT)) and alkaline phosphatase (ALP) below: Not Eligible: AST or ALT > 5xULRR, 1.5xULRR < AST or ALT < 5xULRR and ALP> ULRR, 1xULRR < AST or ALT < 1.5xULRR and ALP> 2.5xULRR, AST or ALT <= ULRR and ALP> 5xULRR For more information please refer to TAXOTERE® (docetaxel) prescribing information

Exclusion Criteria:

* Prior therapy with gefitinib or other EGFR TK inhibitors (HER-1 receptor inhibitors/small molecule or monoclonal antibody therapy)

  * Prior docetaxel treatment for NSCLC
  * Patients with pre-existing peripheral neuropathy ³ grade 2 (NCI CTCAE criteria)
  * Past medical history of interstitial lung disease, drug induced interstitial disease, radiation pneumonitis that required steroid treatment or any evidence of clinically active interstitial lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-10; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Han-Pin Kuo, MD, Principal Investigator — Director of Chest Department, Chang Gung Memorial Hospital, Linkou
Locations (1):
- Research Site, Taipei, Taiwan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 14 patients with locally advanced or metastatic non small cell lung cancer of adenocarcinoma histology previously treated with one platinum based chemotherapy were screened and randomized.
Groups:
- Gefitinib: gefitinib 250mg
- Docetaxel: docetaxel 60mg/m sq
Period: Overall Study
Arm/Group | Gefitinib | Docetaxel
Started | 8 | 6
Completed | 0 | 0
Not Completed | 8 | 6
Not completed — Death | 5 | 1
Not completed — Incorrect enrolment | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Study Termination | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gefitinib | Docetaxel | Total
Number analyzed (Participants) | 8 | 6 | 14
Age Continuous [Mean (Standard Deviation); unit: years] | 67.43 (8.15) | 54.52 (12.34) | 61.89 (11.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 4 | 3 | 7
WHO performance status [Number; unit: participants]
  Normal activity | 0 | 1 | 1
  Restricted activity | 8 | 4 | 12
  In bed less than or equal to 50% of time | 0 | 1 | 1
  In bed more than 50% of the time | 0 | 0 | 0
  100% bedridden | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 60.51 (10.35) | 60.03 (6.4) | 60.31 (8.57)
Height [Mean (Standard Deviation); unit: cm] | 159.3 (7.26) | 162.77 (7.32) | 160.79 (7.22)
BMI [Mean (Standard Deviation); unit: kg/m2] | 23.84 (3.85) | 22.77 (3.27) | 23.39 (3.52)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Event (AE)
Time Frame: From time consent was given to 28 days after last dose of study drug.
Population: Evaluable for Safety population: All patients who recived at least one dose of study drug
Measure: Number; unit: Participants
Arm/Group | Gefitinib | Docetaxel
Number analyzed (Participants) | 8 | 6
Participants | 8 | 6

2. Primary Outcome: Number of Patients With Serious Adverse Events (SAEs)
Time Frame: From time consent was given to 28 days after last dose
Measure: Number; unit: participants
Arm/Group | Gefitinib | Docetaxel
Number analyzed (Participants) | 8 | 6
participants | 2 | 1

ADVERSE EVENTS:
Time Frame: From time consent was given to 28 days after last dose of study drug
Description: Adverse event iformtaion was collectde at each study visit by Information volunteered by the patient, or the patient's care giver; open-ended and non-leading verbal questioning of the patient; and observation by the investigational team, other care providers or relatives.
Arm/Group | Gefitinib | Docetaxel
Serious Adverse Events (participants affected / at risk) | 2/8 | 1/6
Other Adverse Events (participants affected / at risk) | 8/8 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gefitinib (N=8) | Docetaxel (N=6)
Pneumonia (Infections and infestations) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Glaucoma (Eye disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gefitinib (N=8) | Docetaxel (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Borderline glaucoma (Eye disorders) | 1 | 0
Iridocyclitis (Eye disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 2
Asthenia (General disorders) | 0 | 1
Chest discomfort (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 1
Pyrexia (General disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Catheter site infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Wound complication (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 3
Hypoaesthesia (Nervous system disorders) | 1 | 1
Paraplegia (Nervous system disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Bladder disorder (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
This study was terminated early because the purpose of this study had been fulfilled by other supporting data, and due to small number of patients enrolled (14 patients).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No